CLINICAL TRIAL: NCT00671788
Title: A Phase II Evaluation of Dasatinib (Sprycel®, NSC #732517) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170M; NCI-2011-03824 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000594930; GOG-0170M (Other: Gynecologic Oncology Group); GOG-0170M (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2008-05-02; First posted 2008-05-05 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Dasatinib

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive oral dasatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Dasatinib — Given orally
  Other Names: BMS-354825; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well dasatinib works in treating patients with persistent or recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial) in patients with persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events as assessed by CTCAE v3.0.

II. To determine the duration of progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. Objectives in formalin-fixed and paraffin-embedded (FFPE) tumor tissue before treatment with dasatinib.

II. Explore the association between the expression and phosphorylation of biomarkers involved in Src signaling pathways and measures of clinical outcome as well as disease status.

III. Bank residual FFPE tumor tissue for the development and characterization of predictive and/or prognostic biomarkers or the validation of thereapeutic targets.

IV. Objectives in blood drawn before and/or during treatment with dasatinib. V. Isolate, enumerate and characterize circulating tumor cells (CTC) as well as circulating endothelial cells (CEC)/circulating endothelial precursors (CEP).

VI. Prepare a buffy-coat specimen from residual blood remaining after isolation of CTC and CEC/CEP.

VII. Explore whether CTC and CEC/CEP counts or characteristics are associated with measures of clinical outcome and disease status.

VIII. Explore whether the expression and phosphorylation of biomarkers involved in Src signaling pathways in CTC and CEC/CEP are associated with measures of clinical outcome and disease status.

IX. Explore the associations between germline single nucleotide polymorphisms (SNPs) in genes involved in drug metabolism, resistance and DNA repair and measures of clinical outcome and disease status.

X. Bank residual DNA and buffy-coat specimens for the development and characterization of predictive and/or prognostic biomarkers or the validation of therapeutic targets.

XI. Objectives in plasma prepared from blood drawn before and/or during treatment with dasatinib.

XII. Explore the association between angiogenic markers and cytokines including VEGF and measures of clinical outcome and disease status.

XIII. Explore the association between measures of cell-free DNA and measures of clinical outcome and disease status.

XIV. Bank residual plasma for the development and characterization of predictive and/or prognostic biomarkers or the validation of therapeutic targets.

OUTLINE: This is a multicenter study.

Patients receive oral dasatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* All patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or >= 10 mm when measured by spiral CT
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority GOG protocol, if one exists; in general, this would refer to any active GOG Phase III protocol for the same patient population
* Patients who have received one prior regimen must have a GOG Performance Status of 0, 1, or 2; patients who have received two prior regimens must have a GOG Performance Status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated UTI).
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration; six weeks for patient previously treated with monoclonal antibodies
* Prior therapy

  * Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment
  * Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

    * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
    * Note: patients on this non-cytotoxic study are allowed to receive additional cytotoxic chemotherapy for management of recurrent or persistent disease, as defined above
  * Patients must have NOT received any non-cytotoxic therapy for management of recurrent or persistent disease; patients are allowed to receive, but are not required to receive, biologic (non-cytotoxic) therapy as part of their primary treatment regimen
  * Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to CTCAE v 3.0 grade 1
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin greater than or equal to 10 g/dL
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v3.0 grade 1
* Bilirubin less than or equal to 1.5 x ULN, CTCAE v3.0 grade 1
* SGOT and alkaline phosphatase less than or equal to 2.5 x ULN, CTCAE v3.0 grade 1
* Mg++, CA++, phosphate, K+, Na corrected to WNL
* PT/INR, PTT less than or equal to 1 - 1.5 x ULN, CTCAE v 3.0 grade 1 except for patients on therapeutic anticoagulation
* Neuropathy (sensory and motor) less than or equal to CTCAE v 3.0 grade 1
* QTc interval on electrocardiogram must be less than or equal to 450 msec
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements as specified in section 7.0
* Patients of childbearing potential must have a negative serum pregnancy test within 72 hours prior to initiating protocol therapy and be practicing an effective form of contraception during protocol therapy and for at least 4 weeks following completion of protocol therapy
* Patients must not be receiving any other investigational agent
* Patients must be able to swallow whole pills

Exclusion Criteria:

* Patients who have had previous treatment with dasatinib
* Patients who have received radiation to more than 25% of marrow-bearing areas
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last five years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients cannot take St. John's Wort or drink grapefruit juice while on study treatment (discontinue St. John's Wort at least five days before starting dasatinib)
* Patients receiving IV bisphosphonates agree that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia, and may be restarted only if any hypocalcemia has been corrected
* Patients who have a history of cardiac disease:

  * Uncontrolled angina, congestive heart failure (CHF) or myocardial infarction (MI) within six months prior to study entry;
  * Diagnosed congenital long QT syndrome;
  * Clinically significant ventricular arrhythmias (such as ventricular tachycardia [VT], ventricular fibrillation [VF], or Torsades de pointes)
* Patients with hypokalemia or hypomagnesemia if it cannot be corrected to within normal limits prior to dasatinib treatment
* Patients who have a history of significant bleeding disorder unrelated to cancer including:

  * Bleeding diathesis, congenital or acquired within one year prior to initiating protocol therapy (e.g., von Willebrand's disease, acquired anti-factor VIII antibodies);
  * Significant GI bleeding within three months prior to initiating protocol therapy
* Dasatinib is metabolized primarily by the CYP3A4 liver enzyme; consideration should be given to using alternative medications not impacting CYP3A4 while on dasatinib therapy

  * Patients may not be receiving any prohibited potent CYP3A4 inhibitors; for these drugs, a wash-out period of >= 7 days is required prior to starting dasatinib treatment
* Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes; a wash-out period of >= 7 days is required for the following drugs prior to starting dasatinib treatment:

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* The concomitant use of H2 blockers and proton pump inhibitors (PPIs) with dasatinib is not recommended (e.g., famotidine, omeprazole); the use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy; if antacid therapy is needed, the antacid dose should be administered two hours before or after the dose of dasatinib
* Therapeutic anticoagulation is not contraindicated, but for those patients on therapeutic anticoagulation, alteration in coagulation parameters is expected following initiation of dasatinib. For patients on therapeutic anticoagulation, coagulation parameters should be assessed weekly for the first cycle following initiation of dasatinib, weekly for the first cycle following a dose reduction, and weekly for a minimum of two weeks after stopping dasatinib.

Warfarin is permitted for prophylaxis or treatment of thrombosis

* Note: Low molecular weight heparin is permitted provided the patient's PT/INR is =< 1.5; for patients on anticoagulation, coagulation parameters should be assessed weekly for the first cycle following initiation of dasatinib, weekly for the first cycle following a dose reduction, and weekly for a minimum of two weeks after stopping dasatinib

  * Pregnant or nursing women; women of childbearing potential unless using effective contraception as determined by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schilder, Principal Investigator — Gynecologic Oncology Group
Locations (20):
- United States (20):
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 6/2/2008 and closed to accrual on 4/12/2010.
Groups:
- Dasatinib: Dasatinib 100 mg orally once daily every day continuously (one cycle = 28 days) until disease progression or adverse effects prohibit further therapy. If the patient does not experience any side effects when taking this dose of dasatinib for the first cycle of treatment, the dosage will be increased before starting the second cycle of treatment to 140 mg of dasatinib orally, 70 mg in the morning and 70 mg in the evening
Period: Overall Study
Arm/Group | Dasatinib
Started | 35
Completed | 21 (Patients treated until disease progression; completed defined as off treatment due to progression.)
Not Completed | 14
Not completed — Adverse Event | 8
Not completed — Refused further treatment | 3
Not completed — Ineligible | 1
Not completed — MD Decision | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
Age, Customized [Number; unit: participants]
  40-49 years | 4
  50-59 years | 9
  60-69 years | 13
  70-79 years | 6
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since study entry, or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
  CT scan or MRI is used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: Scans to assess progression were done every other cycle for the first 6 months; every three months thereafter; and any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
percentage of participants | 20.6 [10.1 to 35.2]

2. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Per RECIST v1.0 for target lesions and assessed by MRIor CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  CT scan or MRI is used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: Every other cycle for the first 6 months; every three months thereafter; and any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease.
Population: Eligible and treated participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
percentage of participants | 0 [0 to 8.4]

3. Secondary Outcome: Frequency and Severity of Adverse Events as Assessed by CTCAE v3.0
Time Frame: Every cycle during treatment
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free Survival
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
months | 2.1 [1.9 to 3.2]

5. Secondary Outcome: Overall Survival
Time Frame: Every other cycle up to 5 years
Population: Eligible and treated participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
months | 18.4 [12.9 to NA] — NA (not applicable): insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Adverse events were queried for and collected every cycle for the duration of treatment.
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 18/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=34)
Rhinitis (Immune system disorders) | 1
Cardiac General - Other (Cardiac disorders) | 1
Weight Loss (General disorders) | 1
Distention (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1
Cns Ischemia (Nervous system disorders) | 1
Neuropathy-Motor (Nervous system disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=34)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Rhinitis (Immune system disorders) | 3
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 10
Platelets (Blood and lymphatic system disorders) | 6
Leukocytes (Blood and lymphatic system disorders) | 11
Hemoglobin (Blood and lymphatic system disorders) | 31
Prolonged Qtc Interval (Cardiac disorders) | 1
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 2
Ptt (Vascular disorders) | 1
Sweating (General disorders) | 2
Weight Gain (General disorders) | 1
Fever (General disorders) | 3
Weight Loss (General disorders) | 3
Rigors/Chills (General disorders) | 2
Fatigue (General disorders) | 20
Insomnia (General disorders) | 3
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 2
Hot Flashes (Endocrine disorders) | 2
Heartburn (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 3
Taste Alteration (Gastrointestinal disorders) | 4
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Anorexia (Gastrointestinal disorders) | 13
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 10
Hemorrhage, Gu - Vagina (Vascular disorders) | 2
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage, Cns (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 2
Edema: Head And Neck (Blood and lymphatic system disorders) | 3
Ast (Metabolism and nutrition disorders) | 5
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alt (Metabolism and nutrition disorders) | 3
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 2
Mood Alteration - Anxiety (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Neuropathy-Sensory (Nervous system disorders) | 4
Blurred Vision (Eye disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Head/Headache (General disorders) | 7
Pain: Extremity-Limb (General disorders) | 1
Pain: Joint (General disorders) | 4
Pain: Abdominal Pain Nos (General disorders) | 12
Pain: Muscle (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Urinary Retention (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No